CLINICAL TRIAL: NCT06445218
Title: Observational Study of Musculoskeletal Patients in an Emergency Department in France : a Pilot Study
Brief Title: Observational Study of Musculoskeletal Patients in an Emergency Department in France
Acronym: SKUAD-P
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Collaborators: University of Brighton (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0823
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Musculoskeletal Pain
Keywords: Emergency department; musculoskeletal disorder
MeSH Terms: conditions — Musculoskeletal Pain; Emergencies; Musculoskeletal Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data collection: Collection of various data from patients' medical file, such as demographic data, diagnostic results, discharge, treatment....
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Collection of various data from patients' medical file, such as demographic data, diagnostic results, discharge, treatment....

SUMMARY:
The purpose of this study is to estimate the number of patients who come to the emergency department with a musculoskeletal referral, to describe the different types of diagnosis for these patients and their treatment and discharge.

DETAILED DESCRIPTION:
There is a crisis in the emergency department (ED) in France, as their number of consultations have constantly increased over the past ten years . Musculoskeletal disorders (MSK) are the most common cause of consultations in ED, as an example there is an average of 30% of ED consultations being for traumatic issues . Moreover, 90% of all patients coming in ED in France have a favourable prognosis of evolution (no risk of seriousness). In this situation, one of the propositions to help to reduce the ED burden is to allow a direct access to physiotherapists. They are the recommended profession to treat patients for musculoskeletal conditions and several studies showed physiotherapy assessment and treatment in an emergency service is safe and beneficial both for the patients and the hospital teams. They have reported to increase satisfaction, to reduce medications and requirement for expensive imaging on one hand, and to reduce the costs and to give more time to the medical team on the other hand This role does not exist yet in France, although more than 48 countries across the world have implemented it, and French physiotherapists are advocating for it. A recent text has been adopted by the French government allowing patients with recent ankle sprain or low back pain to self-refer to physiotherapists working in hospitals or in care home. . However, this access is very restricted, which will make the implementation difficult as it might not be sufficient to assist the ED. Moreover, there is a lack of information on the number and the type of diagnostic of patients with a MSK label coming to the ED, which makes it difficult to assess the impact this role could have on French ED.

In this context, a retrospective survey, describing how many patients with a musculoskeletal label are coming to the ED, and how they are managed, could help to estimate the worthiness of physiotherapist direct access in French ED.

Question : What is the proportion, the type of diagnostic and the management of musculoskeletal disorder in emergency department in one hospital in France?

ELIGIBILITY:
Inclusion Criteria :

* Patients aged between 18 and 68
* Patients admitted to emergency with a triage by the Reception and Referral Nurse of 0, 1 or 2
* Patients who consulted for one of the following reasons:

Lower limb pain (T13.9) Lower limb trauma (M79.61) Upper limb pain (T11.9) Upper limb trauma (M79.60) Spinal pain (M54.9) Lumbar or flank pain (R10.3) Diffuse/unspecific pain (R52.9) Loss of sensitivity/paraesthesia

- Patients informed of the study and who did not object

Exclusion Criteria :

* Patients with another reason for consultation associated with the first
* Patients under guardianship / curatorship and patients under safeguard of justice.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from musculoskeletal disorders in an emergency department
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Description of the population (diagnoses and treatment) considered to have a potential musculoskeletal disorder after nursing triage | At the end of the study, an average of 3 month
  The description of the patients, triaged by the emergency reception and referral nurse as having a potential musculoskeletal pathology, will be carried out by collecting the different types of diagnoses, based on the International Classification of Diseases - 10th revision (ICD10) and their severity, as well as their age and gender, and the treatments that have been prescribed (medication, imaging, physiotherapy, other…).

SECONDARY OUTCOMES:
Description of the management of patients (duration) with a potential musculoskeletal disorder after nursing triage | At the end of the study, an average of 3 month
  Collection of the duration of care (from registration at the emergency department to the patient's discharge)
Description of the management of patients (number of patients per day of the week) with a potential musculoskeletal disorder after nursing triage | At the end of the study, an average of 3 month
  Collection of the number of patients per day of the week (Monday to Sunday) and by time slots between 8am and 8pm during the day and between 8pm and 8am at night
Description of the management of patients (end-of-care orientation) with a potential musculoskeletal disorder after nursing triage | At the end of the study, an average of 3 month
  Collection of different referrals (hospitalization, return home..) at the end of patient care
Assessment of the prevalence of people with a potential musculoskeletal disorder after nursing triage | At the end of the study, an average of 3 month
  Number of patients with a potential musculoskeletal disorder, after nursing triage, out of the total number of people consulting during the same period

CONTACTS AND LOCATIONS:
Overall Officials: Benoit ANCEL, Principal Investigator — Hôpital NOVO
Locations (1):
- Emergency Service - Hôpital NOVO - Pontoise site, Pontoise, France

REFERENCES:
- [Background] Babatunde OO, Bishop A, Cottrell E, Jordan JL, Corp N, Humphries K, Hadley-Barrows T, Huntley AL, van der Windt DA. A systematic review and evidence synthesis of non-medical triage, self-referral and direct access services for patients with musculoskeletal pain. PLoS One. 2020 Jul 6;15(7):e0235364. doi: 10.1371/journal.pone.0235364. eCollection 2020. PMID 32628696
- [Background] Demont A, Quentin J, Bourmaud A. [Impact of models of care integrating direct access to physiotherapy in primary care and emergency care contexts in patients with musculoskeletal disorders: A narrative review]. Rev Epidemiol Sante Publique. 2020 Sep;68(5):306-313. doi: 10.1016/j.respe.2020.08.001. Epub 2020 Sep 3. French. PMID 32893028
- [Background] Demont A, Bourmaud A, Kechichian A, Desmeules F. The impact of direct access physiotherapy compared to primary care physician led usual care for patients with musculoskeletal disorders: a systematic review of the literature. Disabil Rehabil. 2021 Jun;43(12):1637-1648. doi: 10.1080/09638288.2019.1674388. Epub 2019 Oct 11. PMID 31603709